CLINICAL TRIAL: NCT03372200
Title: Febuxostat-Controlled, Double-Blind, Comparative Study of FYU-981 for Hyperuricemia With or Without Gout to Evaluate the Safety and Noninferiority of FYU-981 (Phase III Study)
Brief Title: Febuxostat-Controlled, Double-Blind, Comparative Study of FYU-981 in Hyperuricemia With or Without Gout
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mochida Pharmaceutical Company, Ltd. (Industry)
Collaborators: Fuji Yakuhin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FYU-981-014
Record Dates: First submitted 2017-12-10; First posted 2017-12-13 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Hyperuricemia With or Without Gout
MeSH Terms: interventions — dotinurad; Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FYU-981 (Experimental)
  Interventions: Drug: FYU-981
- Febuxostat (Active Comparator)
  Interventions: Drug: Febuxostat

INTERVENTIONS:
Drug: FYU-981 — Oral daily dosing for 14 weeks
  Arms: FYU-981
Drug: Febuxostat — Oral daily dosing for 14 weeks
  Arms: Febuxostat

SUMMARY:
FYU-981 or Febuxostat are administrated to hyperuricemia patients (underexcretion and mixed types) with or without gout for 14 weeks to compare the efficacy and safety of these drugs by the method of multicenter, randomized, double-blind, ascending dose regimen.

ELIGIBILITY:
Inclusion Criteria:

* Serum urate level:

  * >= 7.0mg/dL in patients with gouty nodule or with history of gout, or >= 8.0mg/dL in patients with hypertension, diabetes or metabolic syndrome, or >= 9.0mg/dL
* Disease type in the classification of hyperuricemia: Uric acid-underexcretion type or mixed type
* Outpatients

Exclusion Criteria:

* Gouty arthritis within 14 days before randomized allocation
* Secondary hyperuricemia
* HbA1c: >= 8.4%
* Clinically significant cardiac, hepatic, renal, hematologic or endocrine disease
* Kidney calculi or clinically significant urinary calculi
* AST: >= 100 IU/L or ALT: >= 100 IU/L
* eGFR: < 30 mL/min/1.73m^2
* Systolic blood pressure: >= 180 mmHg or diastolic blood pressure: >= 110 mmHg

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Percent reduction from baseline in serum urate level at the final visit | 14 weeks
  Percent reduction from baseline in serum urate level at the final visit

CONTACTS AND LOCATIONS:
Overall Officials: Kazuki Furuno, Study Director — Clinical Research Department
Locations (1):
- Mochida Investigational sites, Tokyo, Japan